CLINICAL TRIAL: NCT02078882
Title: Abatacept For The Treatment Of Primary Biliary Cirrhosis With An Incomplete Biochemical Response To Ursodeoxycholic Acid
Brief Title: Study of Abatacept (Orencia) to Treat Primary Biliary Cirrhosis
Acronym: PBC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christopher Bowlus, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Christopher Bowlus, MD, Professor, Gastroenterology and Hepatology, Internal Medicine, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 599969; IM101-457 (Other: Other)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis; Ursodeoxycholic acid; Abatacept; Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4)
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept 125 mg weekly (Experimental): Open label treatment with Abatacept
  Interventions: Biological: abatacept

INTERVENTIONS:
Biological: abatacept — 125 mg subcutaneously each week for 24 weeks
  Other Names: Orencia

SUMMARY:
The purpose of this study is to determine if abatacept (Orencia) is effective in patients with primary biliary cirrhosis who do not respond adequately to standard treatment with ursodeoxycholic acid (UDCA, Urso, Ursodiol, Actigall).

DETAILED DESCRIPTION:
This is an open label, active treatment trial to assess the efficacy and safety of abatacept in subject with PBC who have had an incomplete biochemical response to UDCA. In this trial, 20 subjects with PBC who have had an incomplete biochemical response to UDCA will be assigned to treatment with weekly subcutaneous injections of 125 mg of abatacept. The treatment phase of the study will last 24 weeks with an off-treatment follow up at Week 36.

Inclusion criteria include:

* Confirmed diagnosis of PBC
* Alkaline phosphatase > 1.67 times the upper limit of normal after 6 months of treatment with UDCA

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PBC diagnosis based upon at least 2 of 3 criteria

  1. Anti-mitochondrial antibody (AMA) titer > 1:40
  2. Alkaline phosphatase > 1.5 times the upper limit of normal for at least 6 months
  3. Liver biopsy findings consistent with PBC
* Incomplete response to UDCA defined by an alkaline phosphatase > 1.67 X the upper limit of normal after 6 months of UDCA at a minimum dose of 13 mg/kg/d
* Taking a stable dose of UDCA for at least 3 months prior to Day 0
* aspartate aminotransferase (AST) and alanine aminotransferase ALT < 5 times the upper limit of normal

Exclusion Criteria:

* Presence of concomitant liver diseases including viral hepatitis, primary sclerosing cholangitis, alcoholic liver disease, Wilson's disease, hemochromatosis, or Gilbert's syndrome.
* Prior liver transplantation
* Decompensated liver disease
* Use of immunosuppressants within 6 months of Day 0
* Use of biologic agents within 12 months of Day 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Bowlus, MD, Principal Investigator — University of California, Davis; M. Eric Gershwin, MD, Principal Investigator — University of California, Davis
Locations (1):
- Univeristy of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: PBC Patient Organization — http://www.pbcers.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept 125 mg Weekly
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 52 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response
Description: Number of Participants with a decrease of alkaline phosphatase by > 40%of the Day 0 level at 24 weeks of treatment.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
Participants | 1

2. Secondary Outcome: Drug Safety
Description: Number of participants with any adverse events, clinically significant changes in vital signs, laboratory test abnormalities, and clinical tolerability of the drug.
Time Frame: Weeks 2, 4, 12, 24, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
Participants | 4

3. Secondary Outcome: Absolute Change in Alkaline Phosphatase
Description: The absolute change in alkaline phosphatase from Day 0 to Week 24.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
IU/L | -2.8 [-97.5 to 42.0]

4. Secondary Outcome: Absolute Change in Alanine Transferase (ALT)
Description: The absolute change in alanine transferase (ALT) from Day 0 to Week 24.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
IU/L | 0.5 [-13.5 to 4.5]

5. Secondary Outcome: Liver Stiffness Measured by Magnetic Resonance Elastography
Description: Change in liver stiffness measured by magnetic resonance elastography from Day 0 to Week 24.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
kPa | -0.1 [-0.43 to 0.20]

6. Secondary Outcome: Primary Billiary Cholangitis Quality of Life
Description: Change in quality of life measured by change in primary biliary cholangitis (PBC)-40 from Day 0 to Week 24. is a patient-derived, disease specific quality of life measure developed and validated for use in PBC with subscores for domains of symptoms, itch, fatigue, cognition, social, and emotional. Subdomains are summed with a total score range of 36 to 200. Higher scores indicate worse quality of life.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
units on a scale | 0 [-4 to 13]

7. Secondary Outcome: Percent Change in Alkaline Phosphatase
Description: The percent change in alkaline phosphatase from Day 0 to Week 24.
Time Frame: Week 24
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
percent change | 0.01 [-0.28 to 0.13]

8. Secondary Outcome: Percent Change in Alanine Transferase (ALT)
Description: The percent change in alanine transferase (ALT) from Day 0 to Week 24.
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
percent change | 0.01 [-0.29 to 0.11]

9. Other Pre Specified Outcome: Immunoglobulin M (IgM) Levels
Description: Change in IgM level from Day 0 to Week 24
Time Frame: Week 24
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Abatacept 125 mg Weekly
Number analyzed (Participants) | 16
mg/dL | 0.0 [-44.0 to 45.0]

10. Other Pre Specified Outcome: Memory T Cell Frequencies
Description: Change in cluster of differentiation 4 (CD4)+ cluster of differentiation 44 (CD44)+ cluster of differentiation 62 ligand (CD62L)- and cluster of differentiation 8+ CD44+ CD62L- frequencies in peripheral blood mononuclear cells from Day 0 to Week 24
Time Frame: Week 24
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Abatacept Levels
Description: Trough serum levels of abatacept
Time Frame: Day 0 and Weeks 4, 12, 24, and 36
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: Adverse events were summarized according to MedDRA System Organ class, MedDRA preferred term, severity and causal relationship assessed by investigators and were reviewed by Data Monitoring Board.
Arm/Group | Abatacept 125 mg Weekly
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept 125 mg Weekly (N=16)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Elevated liver enzymes (Gastrointestinal disorders) | 1 (1)
Right upper quadrant pain (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary Tract Infections (Infections and infestations) | 1 (1)
Urticarial Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Hilar Adenopathy (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02078882/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02078882/ICF_001.pdf